CLINICAL TRIAL: NCT06535490
Title: Prevention of Infection After EUS-FNA of Pancreatic Cystic Lesions: A French Multicenter Prospective Comparative Observational Study
Brief Title: Antibiotic Prophylaxis for EUS-FNA of Pancreatic Cystic Lesions
Acronym: PrePaCyst
Status: Not yet recruiting | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, David KARSENTI, Medical doctor, Principal Investigator, Société Française d'Endoscopie Digestive
Other Study IDs: SFED-165
Record Dates: First submitted 2024-07-28; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cystic Lesion
Keywords: EUS-FNA; Pancreatic cystic lesion; Antibiotic prophylaxis
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Antibiotic Prophylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EUS-FNA for PCL with ATBp: Patients undergoing EUS-FNA for pancreatic cystic lesions WITH ATBp
  Interventions: Procedure: EUS-FNA; Drug: ATBp
- EUS-FNA for PCL without ATBp: Patients undergoing EUS-FNA for pancreatic cystic lesions without ATBp
  Interventions: Procedure: EUS-FNA

INTERVENTIONS:
Procedure: EUS-FNA — Puncture of pancreatic cystic lesion with a fine needle under EUS guidance
  Other Names: EUS fine needle aspiration
Drug: ATBp — Antibiotic prophylaxis consists of a single intravenous administration before or at the beginning of the procedure according to the common practices of each practitioner or unit
  Other Names: Antibiotic prophylaxis
  Groups: EUS-FNA for PCL with ATBp

SUMMARY:
Large prospective comparative observational study in numerous reference centers in France, comparing infectious complications in patients admitted for pancreatic cystic lesions (PCL) aspiration performed with or without antibiotic prophylaxis (ATBp) according to the usual practices.

This is a prospective, comparative, observational, multicenter study, with the primary objective of comparing the infection rates in pancreatic cystic lesions (PCL) aspirated under EUS, with and without the administration of ATBp.

A sample size of 1702 patients will be needed over a 3-year study period.

DETAILED DESCRIPTION:
The complication rate after EUS fine needle aspiration (EUS-FNA) for pancreatic cystic lesions (PCL) is low, around 1-3% according to various series. However, it has long been recommended to perform this procedure under antibiotic prophylaxis (ATBp). Due to the risk of developing resistance to certain classes of antibiotics and the risk of complications, particularly allergic reactions, the role of ATBp in this indication needs to be reconsidered. The latest recommendations from European and French societies do not support the systematic formal indication of ATBp for aspiration under EUS. Because the literature on the subject is sparse and equivocal, practices remain varied (some performing PCL aspirations with and others without ATBp), and scientific societies do not provide a formal stance on the benefit of such ATBp. Therefore, we decided to conduct a very large prospective comparative observational study in numerous reference centers in France (centers of the Research and Action Group in Endoscopy - GRAPHE), comparing infectious complications in patients admitted for EUS-FNA for PCL performed with or without ATBp according to the usual practices .

This is a prospective, comparative, observational, multicenter study.

Primary objective:

Comparison of infection rates after EUS-FNA for pancreatic cystic lesions (PCL) , with and without the administration of ATBp.

Secondary objectives:

Rates of other infectious complications (pulmonary, urinary, etc.) Rates of post-ATBp complications, particularly allergic reactions Prolongation of scheduled hospitalization Evaluation of factors associated with post-EUS aspiration infection of PCL

After the endoscopic exploration, the patient will be monitored for the potential occurrence of complications related to EUS (perforation, hemorrhage, infection, allergy, etc.). Any adverse events will be recorded at 30 days post-procedure.

A sample size of 1702 patients will be needed over a 3-year study period.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for diagnostic aspiration of a pancreatic cystic lesion
* Patient aged 18 years or older
* Patient with ASA 1, ASA 2, ASA 3 status
* No participation in another concurrent clinical study

Exclusion Criteria:

* Patient under 18 years old
* Patient with ASA 4 or ASA 5 status
* Pregnant woman
* Patient with coagulation disorders preventing the performance of an EUS-FNA: PT < 50%, platelets < 50,000/mm³, current effective anticoagulation, ongoing clopidogrel, prasugrel, or ticagrelor treatment
* Patient unable to personally express non-opposition or legally protected adult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic cystic lesions for whom an EUS-FNA is indicated
Sampling Method: Non-Probability Sample
Enrollment: 1702 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Post EUS-FNA PCL infection rate | 30 days
  Post-EUS-FNA infection rate of PCL (patients exhibiting clinical and biological signs - fever >38.5°C, neutrophilic leukocytosis, elevated CRP, pathogen identification in blood cultures - indicative of sepsis requiring prolonged antibiotic therapy). The occurrence of the aforementioned clinical and biological signs, along with imaging evidence (such as cyst wall thickening or presence of intracystic air images) and the absence of another infection source (urinary, pulmonary, venous, etc.) will lead to the diagnosis of post-FNA infection. Centralized validation of infection cases will be conducted by an expert panel based on clinical, biological, and imaging findings.

SECONDARY OUTCOMES:
Rate of urinary infectious complications | 30 days
  Number of patients with at least one urinary infection within 21-30 days after EUS-FNA
Rate of post-ATBp allergic reactions | 30 days
  Number of patients with at least one allergic reaction within 21-30 days after EUS-FNA
Duration and extension of hospitalization | 30 days
  Number of hospitalization days per stay within 30 days following EUS-FNA
Diameter of the needle used for EUS-FNA | 1 days
  25G, 22G, 20G, or 19G
Associated procedures (confocal endomicroscopy or intracystic biopsy) | 1 days
  Yes or No
Appearance of the fluid | 1 day
  Thin, thick, hemorrhagic
Complete aspiration of the cyst fluid | 1 day
  Yes or No
Nature of the PCL | 30 days
  mucinous vs. non-mucinous
Age | 1 day
  Years
Gender | 1 day
  Male or female
Diabetes | 1 day
  Yes or No
Immunosuppression | 1 day
  Yes or No
BMI | 1 day
  Weight/(size)2 expressed in in kg/m^2
history of aspiration of the same lesion | 1 day
  Yes or No
Rate of pulmonary infectious complications | 30 days
  Number of patients with at least one pulmonary infection within 21-30 days after EUS-FNA

CONTACTS AND LOCATIONS:
Overall Officials: David KARSENTI, Study Chair — Societe Française d'Endoscopie Digestive
Locations (1):
- Clinique Paris-Bercy, Charenton-le-Pont, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Polkowski M, Jenssen C, Kaye P, Carrara S, Deprez P, Gines A, Fernandez-Esparrach G, Eisendrath P, Aithal GP, Arcidiacono P, Barthet M, Bastos P, Fornelli A, Napoleon B, Iglesias-Garcia J, Seicean A, Larghi A, Hassan C, van Hooft JE, Dumonceau JM. Technical aspects of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Technical Guideline - March 2017. Endoscopy. 2017 Oct;49(10):989-1006. doi: 10.1055/s-0043-119219. Epub 2017 Sep 12. PMID 28898917
- [Result] Facciorusso A, Mohan BP, Tacelli M, Crino SF, Antonini F, Fantin A, Barresi L. Use of antibiotic prophylaxis is not needed for endoscopic ultrasound-guided fine-needle aspiration of pancreatic cysts: a meta-analysis. Expert Rev Gastroenterol Hepatol. 2020 Oct;14(10):999-1005. doi: 10.1080/17474124.2020.1797486. Epub 2020 Jul 25. PMID 32674699
- [Result] Facciorusso A, Arevalo-Mora M, Conti Bellocchi MC, Bernardoni L, Ramai D, Gkolfakis P, Loizzi D, Muscatiello N, Ambrosi A, Tartaglia N, Robles-Medranda C, Stasi E, Ofosu A, Crino SF. Impact of Antibiotic Prophylaxis on Infection Rate after Endoscopic Ultrasound Through-the-Needle Biopsy of Pancreatic Cysts: A Propensity Score-Matched Study. Diagnostics (Basel). 2022 Jan 16;12(1):211. doi: 10.3390/diagnostics12010211. PMID 35054378
- [Result] Facciorusso A, Buccino VR, Turco A, Antonino M, Muscatiello N. Antibiotics Do Not Decrease the Rate of Infection After Endoscopic Ultrasound Fine-Needle Aspiration of Pancreatic Cysts. Dig Dis Sci. 2019 Aug;64(8):2308-2315. doi: 10.1007/s10620-019-05655-x. Epub 2019 May 7. PMID 31065897
- [Result] Klein A, Qi R, Nagubandi S, Lee E, Kwan V. Single-dose intra-procedural ceftriaxone during endoscopic ultrasound fine-needle aspiration of pancreatic cysts is safe and effective: results from a single tertiary center. Ann Gastroenterol. 2017;30(2):237-241. doi: 10.20524/aog.2016.0118. Epub 2016 Dec 22. PMID 28243046
- [Result] Guarner-Argente C, Shah P, Buchner A, Ahmad NA, Kochman ML, Ginsberg GG. Use of antimicrobials for EUS-guided FNA of pancreatic cysts: a retrospective, comparative analysis. Gastrointest Endosc. 2011 Jul;74(1):81-6. doi: 10.1016/j.gie.2011.03.1244. PMID 21704808
- [Result] Lee LS, Saltzman JR, Bounds BC, Poneros JM, Brugge WR, Thompson CC. EUS-guided fine needle aspiration of pancreatic cysts: a retrospective analysis of complications and their predictors. Clin Gastroenterol Hepatol. 2005 Mar;3(3):231-6. doi: 10.1016/s1542-3565(04)00618-4. PMID 15765442
- [Result] Colan-Hernandez J, Sendino O, Loras C, Pardo A, Gornals JB, Concepcion M, Sanchez-Montes C, Murzi M, Andujar X, Velasquez-Rodriguez J, Rodriguez de Miguel C, Fernandez-Esparrach G, Gines A, Guarner-Argente C. Antibiotic Prophylaxis Is Not Required for Endoscopic Ultrasonography-Guided Fine-Needle Aspiration of Pancreatic Cystic Lesions, Based on a Randomized Trial. Gastroenterology. 2020 May;158(6):1642-1649.e1. doi: 10.1053/j.gastro.2020.01.025. Epub 2020 Jan 20. PMID 31972236